CLINICAL TRIAL: NCT01895803
Title: To Find Factors That Inhibit Women Who Smoke to do Pap Smear Test
Brief Title: The Factors That Inhibit Women Who Smoke to do Pap Smear Test
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: HYMC 0047-13
Record Dates: First submitted 2013-06-26; First posted 2013-07-11 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-06

CONDITIONS: Smoking Woman; 18-60 Years Old
Keywords: smoking woman

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- smoking woman 18-60 years old

SUMMARY:
Discovery of factors affect the decision of the woman to perform or not to perform a Pap test.Participate in the study 100 women who smoke. Age range 18-60

DETAILED DESCRIPTION:
The data collected through questionnaires to the women. Data analysis will be performed by using Statistical Analysis- SPSS

ELIGIBILITY:
Inclusion Criteria:

* smoking woman 18-60 years old

Exclusion Criteria:

* not smoking Not want to participate in the study

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: smoking woman 18-60 years old
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-07; Primary Completion 2013-09 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Why does not a woman who smokes do Pap test | 2 Months
  Discovery of factors affect the decision of the woman to perform or not to perform a Pap test.
  Participate in the study 100 women who smoke. Age range 18-60
  The data collected through questionnaires to the women. Data analysis will be performed by using Statistical Analysis- SPSS

CONTACTS AND LOCATIONS:
Locations (1):
- Afllalo Yael, Hadera, Israel